CLINICAL TRIAL: NCT00619814
Title: Is Barium Enema an Adequate Diagnostic Test for Patients With Positive FOBT?
Acronym: DCBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Caribbean Healthcare System (U.S. Federal Agency)
Responsible Party: Doris Toro, MD
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 00171
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Cancer
Keywords: Colon polyps; Fecal occult blood test; Double contrast barium enema; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort group (Other): Cohort group of asymptomatic patients 50-80 years old with a positive fecal occult blood test done for colorectal cancer screening.
  Interventions: Procedure: Double-contrast Barium enema, colonoscopy

INTERVENTIONS:
Procedure: Double-contrast Barium enema, colonoscopy — This is a blinded cohort study comparing double contrast barium enema (DCBE) and colonoscopy in detecting polyps and/or cancer in patients with positive FOBT. Initial evaluation consisted of complete clinical history and physical examination. A DCBE and a colonoscopy were performed in all patients. All polyps identified during colonoscopy were removed and classified by histology. Sensitivity and specificity of DCBE for polyp and/or cancer detection was determined. Tolerability and grade of satisfaction with study procedures was assessed.

SUMMARY:
The research protocol aim is to compare diagnostic tools for the proper evaluation of patient with fecal occult blood test positive (FOBT +), a routine screening test for colorecatl carcinoma. The purpose of this study is to determine if Double Contrast Barium Enema (DCBE), a specialized radiographic exam of the colon, is a reasonable alternative for the evaluation of patients with positive fecal occult blood as compared to colonoscopy, which is considered the best evaluation method. Colonoscopy involves the direct visualization of the colon using a flexible instrument. This permits the removal of polyps and to obtain biopsies. It involves additional risks, discomfort and costs. In fact the DCBE is the experimental procedure in this protocol.

Additional aims of this study are: to determine the localization, number, size and pathologic characteristics, if applicable, of findings in colonoscopy and/or DCBE and to determine the patient preference between both studies.

This study is limited to those patients 50 years or older who are at average risk for colon cancer and who had a positive fecal occult blood screening test.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients older than 50 years of age, with at least one positive FOBT
* Without history of colon cancer and/or polyps
* Gross gastrointestinal bleeding or prior colonoscopy or DCBE
* Who were willing to participate in the study
* Were included in the investigation.

Exclusion Criteria:

* Patients with poor cardio-respiratory condition
* Coagulation deficiency, use of anticoagulants or other drugs affecting coagulation
* Severe renal or liver disease
* Hospitalized patients and palpable abdominal or rectal mass were excluded from the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)